CLINICAL TRIAL: NCT00423670
Title: A Safety and Efficacy Study of SCH 503034 in Previously Untreated Subjects With Chronic Hepatitis C Infected With Genotype 1
Brief Title: Safety and Efficacy of SCH 503034 in Previously Untreated Subjects With Chronic Hepatitis C Infected With Genotype 1 (Study P03523)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P03523; EudraCT No. 2006-002543-92
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Results first posted 2011-06-15 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Arm 1. PEG +RBV for 48 Wks (Part I) (Active Comparator): Participants treated with PegIntron (1.5 μg/kg, once weekly [QW]) and Ribavirin (800 to 1400 mg/day) for 48 weeks.
  Participants with detectable HCV-RNA levels after 24 weeks of treatment had the option of crossing over to receive 24 weeks of PegIntron (1.5 μg/kg, QW), Ribavirin (800 to 1400 mg/day), and boceprevir (800 mg three times daily [TID]) for 24 additional weeks. The participants that crossed over to receive boceprevir formed Arm 8. The total treatment duration was up to 54 weeks.
  Interventions: Drug: peginterferon-alfa 2b (PegIntron); Drug: ribavirin
- Arm 2. PEG + RBV + BOC for 28 Wks (Part I) (Experimental): Participants receiving boceprevir (800 mg TID) plus PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for up to 28 weeks.
  Interventions: Drug: boceprevir (SCH 503034); Drug: peginterferon-alfa 2b (PegIntron); Drug: ribavirin
- Arm 3. PEG + RBV + BOC (from Wk 4) for 24 Wks (Part I) (Experimental): Participants receiving a lead-in treatment with PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for 4 weeks, followed by boceprevir (800 mg TID) plus PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for up to 24 weeks.
  Interventions: Drug: boceprevir (SCH 503034); Drug: peginterferon-alfa 2b (PegIntron); Drug: ribavirin
- Arm 4. PEG +RBV + BOC for 48 Wks (Part I) (Experimental): Participants receiving boceprevir (800 mg TID) plus PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for up to 48 weeks.
  Interventions: Drug: boceprevir (SCH 503034); Drug: peginterferon-alfa 2b (PegIntron); Drug: ribavirin
- Arm 5. PEG + RBV + BOC (from Wk 4) for 44 Wks (Part I) (Experimental): Participants receiving a lead-in treatment with PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for 4 weeks, followed by boceprevir (800 mg TID) plus PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for up to 44 weeks.
  Interventions: Drug: boceprevir (SCH 503034); Drug: peginterferon-alfa 2b (PegIntron); Drug: ribavirin
- Arm 6. PEG + RBV + BOC for 48 Wks (Part II) (Experimental): Participants receiving PegIntron (1.5 μg/kg QW), ribavirin (800 to 1400 mg/day) and boceprevir (800 mg TID) for up to 48 weeks during Part II of the study. Part II was initiated after participants were fully enrolled for Part I.
  Interventions: Drug: boceprevir (SCH 503034); Drug: peginterferon-alfa 2b (PegIntron); Drug: ribavirin
- Arm 7. PEG +Low-dose RBV + BOC for 48 Wks (Part II) (Experimental): Participants receiving PegIntron (1.5 μg/kg QW), low-dose ribavirin (400 to 1000 mg/day) and boceprevir (800 mg TID) for up to 48 weeks (Arm 7) during Part II of the study. Part II was initiated after participants were fully enrolled for Part I.
  Interventions: Drug: boceprevir (SCH 503034); Drug: peginterferon-alfa 2b (PegIntron); Drug: ribavirin (low-dose)
- Arm 8. PEG + RBV + BOC (from Wk 24) for 48 Wks (Part I) (Experimental): Participants that started in Arm 1 and had detectable HCV-RNA levels after 24 weeks of treatment had the option of receiving boceprevir (800 mg TID) with
  PegIntron (1.5 μg/kg QW), and ribavirin (800 to 1400 mg/day). Participants that took the option of crossing over to receive PegIntron, ribavirin, and boceprevir (800 mg TID) for 24 additional weeks constitute Arm 8. The total treatment duration was up to 54 weeks.
  Interventions: Drug: boceprevir (SCH 503034); Drug: peginterferon-alfa 2b (PegIntron); Drug: ribavirin

INTERVENTIONS:
Drug: boceprevir (SCH 503034) — 200 mg capsules taken as 800 mg orally three times daily (TID)
  Other Names: Boceprevir, Victrelis, SCH 503034
  Arms: Arm 2. PEG + RBV + BOC for 28 Wks (Part I); Arm 3. PEG + RBV + BOC (from Wk 4) for 24 Wks (Part I); Arm 4. PEG +RBV + BOC for 48 Wks (Part I); Arm 5. PEG + RBV + BOC (from Wk 4) for 44 Wks (Part I); Arm 6. PEG + RBV + BOC for 48 Wks (Part II); Arm 7. PEG +Low-dose RBV + BOC for 48 Wks (Part II); Arm 8. PEG + RBV + BOC (from Wk 24) for 48 Wks (Part I)
Drug: peginterferon-alfa 2b (PegIntron) — 1.5 μg/kg subcutaneously (SC) once weekly (QW)
Drug: ribavirin — 200 mg capsules in doses of 800 to 1400 mg/day (based on weight) taken orally divided twice daily
  Arms: Arm 1. PEG +RBV for 48 Wks (Part I); Arm 2. PEG + RBV + BOC for 28 Wks (Part I); Arm 3. PEG + RBV + BOC (from Wk 4) for 24 Wks (Part I); Arm 4. PEG +RBV + BOC for 48 Wks (Part I); Arm 5. PEG + RBV + BOC (from Wk 4) for 44 Wks (Part I); Arm 6. PEG + RBV + BOC for 48 Wks (Part II); Arm 8. PEG + RBV + BOC (from Wk 24) for 48 Wks (Part I)
Drug: ribavirin (low-dose) — 200 mg capsules in doses of 400 to 1000 mg/day (based on weight) taken orally divided twice daily
  Arms: Arm 7. PEG +Low-dose RBV + BOC for 48 Wks (Part II)

SUMMARY:
This was an open-label, randomized safety and efficacy trial in adult, treatment-naïve Chronic Hepatitis C (CHC) participants with genotype 1 infection. The study conducted in 2 parts, compared standard-of-care PegIntron (1.5 μg/kg, once weekly [QW]), plus ribavirin (800 to 1400 mg/day), for 48 weeks to five treatment paradigms containing boceprevir (SCH 503034) 800 mg thrice a day (TID). The five treatments included boceprevir (BOC) plus standard-of-care for 28 or 48 weeks, with and without a 4-week lead-in with PegIntron (PEG) and ribavirin (RBV), and exploration of PegIntron plus low-dose ribavirin (400 to 1000 mg/day) plus boceprevir for 48 weeks.

DETAILED DESCRIPTION:
The study was conducted in 2 parts.

Part 1 of the study had 5 arms using weight based ribavirin 800-1400 mg/day and compared:

* PegIntron and ribavirin for 48 weeks (Arm 1 - Control)
* PegIntron, ribavirin, and boceprevir for 28 weeks (Arm 2)
* Lead-in with PegIntron and ribavirin for 4 weeks followed by PegIntron, ribavirin and boceprevir for 24 weeks (Arm 3)
* PegIntron, ribavirin and boceprevir for 48 weeks (Arm 4)
* Lead-in with PegIntron and ribavirin for 4 weeks, followed by PegIntron, ribavirin and boceprevir for 44 weeks (Arm 5)

Participants from Arm 1 receiving PegIntron and ribavirin that were HCV positive after 24 weeks of treatment had the option to receive boceprevir in combination with PegIntron and ribavirin for an additional 24 weeks. All participants from Arm 1 that started boceprevir after Week 24 formed the crossover arm (Arm 8).

Part 2 of the study assessed the safety and efficacy of low dose ribavirin (400-1000 mg/day) and compared:

* PegIntron, ribavirin (800-1400 mg/day) and boceprevir for 48 weeks (Arm 6)
* PegIntron, low-dose ribavirin (400-1000 mg/day) and boceprevir for 48 weeks (Arm 7)

Follow-up for all participants was up to 72 weeks after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years;
* Body weight between 45 and 125 kg;
* Documented chronic hepatitis C genotype 1;
* Liver biopsy with histology consistent with chronic hepatitis and no other etiology for chronic liver disease within of 5 years of Day 1;
* Participant and participant's partner(s) must each agree to use acceptable methods of contraception 2 weeks prior to Day 1 and at least 6 months after the last dose of study medication;
* Written informed consent.

Exclusion Criteria:

Include, but are not limited to, the following:

* Prior treatment for hepatitis C;
* Co-infection with HIV or hepatitis B virus (HBsAg positive);
* Evidence of decompensated liver disease;
* Diabetic and hypertensive participants with clinically significant ocular exam findings;
* Pre-existing psychiatric condition, including but not limited to:

  * Current moderate or severe depression;
  * History of depression associated with any of the following:

    * Hospitalization for depression;
    * Electroconvulsive therapy for depression;
    * Depression that resulted in a prolonged absence from work and/or significant disruption of daily functions;
  * Suicidal or homicidal ideation and/or attempt;
  * History of severe psychiatric disorders (including but not limited to schizophrenia, psychosis, bipolar disorder, post-traumatic stress disorder or mania);
  * Past history or current use of lithium;
  * Past history or current use of antipsychotic drugs for listed conditions.
* Substance abuse within protocol specified timeframes;
* Pre-existing medical conditions that could interfere with the participant's participation in and completion of the study, including but not limited to chronic pulmonary disease, cardiac dysfunction or immunologically-mediated disease;
* Active or suspected malignancy or history of malignancy within the past 5 years;
* Participants who are pregnant or nursing; participants who intend to become pregnant during the study period. Male participants with partners who are, or intend to become, pregnant during the study period.
* Treatment with any investigational drug or participation in any clinical trial 30 days within Screening;
* Hemoglobin <12 g/dL for females and <13 g/dL for males;
* Neutrophils <1500 mm^3; Blacks: <1200/mm^3;
* Platelets <100,000/mm^3;
* Other clinically significant laboratory test abnormalities.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 765 (Actual)
Dates: Start 2007-01; Primary Completion 2008-08 (Actual); Study Completion 2008-11 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Kwo PY, Lawitz EJ, McCone J, Schiff ER, Vierling JM, Pound D, Davis MN, Galati JS, Gordon SC, Ravendhran N, Rossaro L, Anderson FH, Jacobson IM, Rubin R, Koury K, Pedicone LD, Brass CA, Chaudhri E, Albrecht JK; SPRINT-1 investigators. Efficacy of boceprevir, an NS3 protease inhibitor, in combination with peginterferon alfa-2b and ribavirin in treatment-naive patients with genotype 1 hepatitis C infection (SPRINT-1): an open-label, randomised, multicentre phase 2 trial. Lancet. 2010 Aug 28;376(9742):705-16. doi: 10.1016/S0140-6736(10)60934-8. Epub 2010 Aug 6. PMID 20692693

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 765 participants were screened in the study, 598 were randomized of which 3 participants were not
  treated (Arm 1-7). Participants were assigned to Part I (with standard dosing for ribavirin) or Part II (to explore low-dose ribavirin). All participants that completed or discontinued treatment were scheduled to enter follow-up phase per protocol.
Pre-assignment Details: Participants in Arm 1 (Part I) who had detectable Hepatitis C Virus-ribonucleic acid (HCV-RNA) at Treatment Week (TW) 24 were offered boceprevir in addition to PegIntron and ribavirin for an additional 24 weeks of treatment, and switched to a new arm, Arm 8.
Groups:
- Arm 1. PEG +RBV for 48 Wks (Part I): PegIntron (1.5 μg/kg, once weekly [QW]) plus ribavirin (800 to 1400 mg/day) for 48 weeks.
  • Participants with detectable HCV-RNA levels after 24 weeks of treatment had the option of crossing over to receive 24 weeks of PegIntron, ribavirin, and boceprevir (800 mg, thrice a day [TID]) for 24 additional weeks. Total treatment duration was up to 54 weeks.
- Arm 2. PEG + RBV + BOC for 28 Wks (Part I): Boceprevir (800 mg TID) plus PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for up to 28 weeks.
- Arm 3. PEG + RBV + BOC (From Wk 4) for 24 Wks (Part I): PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for 4 weeks lead-in followed by boceprevir (800 mg TID) plus PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for up to 24 weeks.
- Arm 4. PEG +RBV + BOC for 48 Wks (Part I): Boceprevir (800 mg TID) plus PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for up to 48 weeks.
- Arm 5. PEG + RBV + BOC (From Wk 4) for 44 Wks (Part I): PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for 4 weeks lead-in followed by boceprevir (800 mg TID) plus PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for up to 44 weeks.
- Arm 6. PEG + RBV + BOC for 48 Wks (Part II): PegIntron (1.5 μg/kg QW), ribavirin (800 to 1400 mg/day) and boceprevir (800 mg TID) for up to 48 weeks.
- Arm 7. PEG +Low-dose RBV + BOC for 48 Wks (Part II): PegIntron (1.5 μg/kg QW), ribavirin (400 to 1000 mg/day) and boceprevir (800 mg TID) for up to 48 weeks.
- Arm 8. PEG + RBV + BOC (From Wk 24) for 48 Wks (Part I): Participants that started in Arm 1 and had detectable HCV-RNA levels after 24 weeks of treatment had the option of receiving boceprevir (800 mg TID) with PegIntron (1.5 μg/kg QW), ribavirin (800 to 1400 mg/day). Participants that took the option of crossing over to receive 24 weeks of PegIntron, ribavirin, and boceprevir (800 mg TID) for 24 additional weeks constitute Arm 8. The total treatment duration was up to 54 weeks.
Period: Treatment Period
Arm/Group | Arm 1. PEG +RBV for 48 Wks (Part I) | Arm 2. PEG + RBV + BOC for 28 Wks (Part I) | Arm 3. PEG + RBV + BOC (From Wk 4) for 24 Wks (Part I) | Arm 4. PEG +RBV + BOC for 48 Wks (Part I) | Arm 5. PEG + RBV + BOC (From Wk 4) for 44 Wks (Part I) | Arm 6. PEG + RBV + BOC for 48 Wks (Part II) | Arm 7. PEG +Low-dose RBV + BOC for 48 Wks (Part II) | Arm 8. PEG + RBV + BOC (From Wk 24) for 48 Wks (Part I)
Started | 104 | 107 | 103 | 103 | 103 | 16 | 59 | 36 (Arm 8 were Arm 1 participants that were positive for HCV-RNA at TW 24 and had the option to switch.)
Completed | 52 | 77 | 76 | 63 | 76 | 8 | 28 | 15
Not Completed | 52 | 30 | 27 | 40 | 27 | 8 | 31 | 21
Not completed — Switched to Arm 8 at TW 24 | 36 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 8 | 12 | 15 | 20 | 9 | 4 | 7 | 2
Not completed — Protocol-defined clinical event | 0 | 7 | 4 | 12 | 5 | 4 | 16 | 15
Not completed — Lost to Follow-up | 2 | 1 | 3 | 1 | 6 | 0 | 3 | 1
Not completed — Subject withdrew (not treatment related) | 3 | 9 | 4 | 4 | 5 | 0 | 3 | 0
Not completed — Investigator decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Non-compliance with protocol | 3 | 1 | 1 | 3 | 2 | 0 | 2 | 2
Period: Follow-up Period
Arm/Group | Arm 1. PEG +RBV for 48 Wks (Part I) | Arm 2. PEG + RBV + BOC for 28 Wks (Part I) | Arm 3. PEG + RBV + BOC (From Wk 4) for 24 Wks (Part I) | Arm 4. PEG +RBV + BOC for 48 Wks (Part I) | Arm 5. PEG + RBV + BOC (From Wk 4) for 44 Wks (Part I) | Arm 6. PEG + RBV + BOC for 48 Wks (Part II) | Arm 7. PEG +Low-dose RBV + BOC for 48 Wks (Part II) | Arm 8. PEG + RBV + BOC (From Wk 24) for 48 Wks (Part I)
Started | 97 | 100 | 96 | 96 | 91 | 14 | 50 | 35
Completed | 94 | 84 | 85 | 91 | 89 | 14 | 41 | 32
Not Completed | 3 | 16 | 11 | 5 | 2 | 0 | 9 | 3
Not completed — Lost to Follow-up | 0 | 12 | 8 | 3 | 1 | 0 | 5 | 0
Not completed — Subject withdrew (not treatment related) | 1 | 4 | 2 | 1 | 1 | 0 | 1 | 1
Not completed — Non-compliance with protocol | 2 | 0 | 1 | 1 | 0 | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Arm 1. PEG +RBV for 48 Wks (Part I): PegIntron (1.5 μg/kg QW) plus ribavirin (800 to 1400 mg/day) for 48 weeks.
  • Participants with detectable HCV-RNA levels after 24 weeks of treatment had to receive 24 weeks of PegIntron, ribavirin and boceprevir (800 mg TID) for 24 additional weeks. Total treatment duration was up to 54 weeks.
- Arm 3. PEG + RBV + BOC (From Wk 4) for 24 Wks (Part I): PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for 4 weeks lead in followed by boceprevir (800 mg TID) plus PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for up to 24 weeks.
- Arm 5. PEG + RBV+ BOC (From Wk 4) for 44 Wks (Part I): PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for 4 weeks lead in followed by boceprevir (800 mg TID) plus PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for up to 44 weeks.
- Total: Total of all reporting groups
Arm/Group | Arm 1. PEG +RBV for 48 Wks (Part I) | Arm 2. PEG + RBV + BOC for 28 Wks (Part I) | Arm 3. PEG + RBV + BOC (From Wk 4) for 24 Wks (Part I) | Arm 4. PEG +RBV + BOC for 48 Wks (Part I) | Arm 5. PEG + RBV+ BOC (From Wk 4) for 44 Wks (Part I) | Arm 6. PEG + RBV + BOC for 48 Wks (Part II) | Arm 7. PEG +Low-dose RBV + BOC for 48 Wks (Part II) | Total
Number analyzed (Participants) | 104 | 107 | 103 | 103 | 103 | 16 | 59 | 595
Age, Continuous [Mean (Standard Deviation); unit: years] — Overall age characteristics were displayed for Arm 1 through Arm 7. Participants from Arm 1 (Part I) who had detectable HCV-RNA at TW 24, had the option to switch to a new arm, Arm 8.
  years | 48.3 (6.9) | 46.4 (8.0) | 47.7 (7.4) | 46.7 (8.8) | 47.6 (8.3) | 50.3 (8.5) | 48.7 (5.8) | 47.5 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Overall gender characteristics were displayed for Arm 1 through Arm 7. Participants from Arm 1 (Part I) who had detectable HCV-RNA TW 24, had the option to switch to a new arm, Arm 8.
  Participants
    Female | 34 | 44 | 52 | 40 | 45 | 7 | 18 | 240
    Male | 70 | 63 | 51 | 63 | 58 | 9 | 41 | 355

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Virologic Response (SVR)
Description: Participants with undetectable HCV-RNA at FW 24 up to EOF had achieved SVR.
  Participants missing data at FW 24 were considered to achieve SVR if
  1. he/she had undetectable HCV-RNA at FW 12 or later
  2. he/she returned later to the study center and had undetectable HCV-RNA.
  HCV-RNA in plasma samples was detected with reverse-transcriptase-polymerase chain reaction (RT-PCR) assay, with a lower limit of detection (LLD) of 29 international units/mL (IU/mL).
  A participant in Arm 2 with undetectable HCV-RNA at FW 24 had detectable HCV-RNA after FW 24. He is not considered to achieve SVR.
Time Frame: From follow-up week (FW) 24 up to end of follow-up (EOF)
Population: Intent-to-Treat (ITT) population: All randomized participants who received at least one dose of any study medication (PegIntron, ribavirin, or boceprevir).
Measure: Number; unit: Participants
Arm/Group | Arm 1. PEG +RBV for 48 Wks (Part I) | Arm 2. PEG + RBV + BOC for 28 Wks (Part I) | Arm 3. PEG + RBV + BOC (From Wk 4) for 24 Wks (Part I) | Arm 4. PEG +RBV + BOC for 48 Wks (Part I) | Arm 5. PEG + RBV+ BOC (From Wk 4) for 44 Wks (Part I) | Arm 6. PEG + RBV + BOC for 48 Wks (Part II) | Arm 7. PEG +Low-dose RBV + BOC for 48 Wks (Part II)
Number analyzed (Participants) | 104 | 107 | 103 | 103 | 103 | 16 | 59
Participants | 39 | 58 | 58 | 69 | 77 | 8 | 21
Statistical Analysis 1: Comparison: Arm 1. PEG +RBV for 48 Wks (Part I) vs Arm 2. PEG + RBV + BOC for 28 Wks (Part I); Test type: Superiority or Other; p = 0.0126, Cochran-Mantel Haenszel Chi-square test; Adjusted for baseline stratification factors: black versus non-black, and cirrhosis versus no cirrhosis; Percent difference in SVR = 16.7, 95% CI 2-sided [3.5 to 30]
Statistical Analysis 2: Comparison: Arm 1. PEG +RBV for 48 Wks (Part I) vs Arm 3. PEG + RBV + BOC (From Wk 4) for 24 Wks (Part I); Test type: Superiority or Other; p = 0.0048, Cochran-Mantel Haenszel Chi-square test; Adjusted for baseline stratification factors: black versus non-black, and cirrhosis versus no cirrhosis; Percent difference in SVR = 18.8, 95% CI 2-sided [5.5 to 32.2]
Statistical Analysis 3: Comparison: Arm 1. PEG +RBV for 48 Wks (Part I) vs Arm 4. PEG +RBV + BOC for 48 Wks (Part I); Test type: Superiority or Other; p < 0.0001, Cochran-Mantel Haenszel Chi-square test; Adjusted for baseline stratification factors: black versus non-black, and cirrhosis versus no cirrhosis; Percent difference in SVR = 29.5, 95% CI 2-sided [16.5 to 42.5]
Statistical Analysis 4: Comparison: Arm 1. PEG +RBV for 48 Wks (Part I) vs Arm 5. PEG + RBV+ BOC (From Wk 4) for 44 Wks (Part I); Test type: Superiority or Other; p < 0.0001, Cochran-Mantel Haenszel Chi-square test; Adjusted for baseline stratification factors: black versus non-black, and cirrhosis versus no cirrhosis; Percent difference in SVR = 37.3, 95% CI 2-sided [24.7 to 49.8]

2. Secondary Outcome: Number of Participants With SVR Based on a 4-week lead-in Treatment With PegIntron and Ribavirin
Description: Number of participants with SVR (undetectable plasma HCV-RNA at FW 24 up to EOF). To assess the effect of lead-in treatment on SVR, participants with (Arm 3 and Arm 5) or without (Arm 2 and Arm 4) lead-in were pooled.
  Participants missing data at FW 24 were considered to achieve SVR if
  1. he/she had undetectable HCV-RNA at FW 12 or later
  2. he/she returned later to the study center and had undetectable HCV-RNA.
  HCV-RNA in plasma samples was detected with an RT-PCR assay. The LLD for the assay was 29 IU/mL.
Time Frame: From FW 24 up to EOF
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Arm 3 and Arm 5. PEG + RBV + BOC (From Wk 4): PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for 4 weeks lead in followed by boceprevir (800 mg TID) plus PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for up to 44 weeks.
- Arm 2 and Arm 4. PEG + RBV + BOC: Boceprevir (800 mg TID) plus PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for up to 48 weeks.
Arm/Group | Arm 3 and Arm 5. PEG + RBV + BOC (From Wk 4) | Arm 2 and Arm 4. PEG + RBV + BOC
Number analyzed (Participants) | 206 | 210
Participants | 135 | 127
Statistical Analysis 1: Comparison: Arm 3 and Arm 5. PEG + RBV + BOC (From Wk 4) vs Arm 2 and Arm 4. PEG + RBV + BOC; Test type: Superiority or Other; p = 0.2864, Cochran-Mantel-Haenszel Chi-Square Test; Adjusted for baseline stratification factors: black versus non black, and cirrhosis versus no cirrhosis; Percent difference in SVR rates = 5.1, 95% CI 2-sided [-4.2 to 14.3]

3. Secondary Outcome: Number of Participants With SVR Based on Duration of Boceprevir Treatment
Description: Number of participants with SVR (undetectable plasma HCV-RNA at FW 24 up to EOF). Participants from treatment arms receiving boceprevir for 28-weeks (Arm 2 and Arm 3) were pooled, and those receiving boceprevir for 48-weeks (Arm 4 and Arm 5) were pooled for the analysis.
  Participants missing data at FW 24 were considered to achieve SVR if
  1. he/she had undetectable HCV-RNA at FW 12 or later
  2. he/she returned later to the study center and had undetectable HCV-RNA.
  HCV-RNA in plasma samples was detected with an RT-PCR assay. The LLD for the assay was 29 IU/mL.
Time Frame: From FW 24 up to EOF
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Arm 4 and Arm 5. PEG + RBV + BOC (48 Weeks): PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) with or without a 4 weeks lead with boceprevir (800 mg TID) for 48 weeks.
- Arm 2 and Arm 3. PEG + RBV + BOC (28 Weeks): PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) with or without a 4 weeks lead with boceprevir (800 mg TID) for 28 weeks.
Arm/Group | Arm 4 and Arm 5. PEG + RBV + BOC (48 Weeks) | Arm 2 and Arm 3. PEG + RBV + BOC (28 Weeks)
Number analyzed (Participants) | 206 | 210
Participants | 146 | 116
Statistical Analysis 1: Comparison: Arm 4 and Arm 5. PEG + RBV + BOC (48 Weeks) vs Arm 2 and Arm 3. PEG + RBV + BOC (28 Weeks); Test type: Superiority or Other; p = 0.0009, Cochran-Mantel-Haenszel Chi-Square Test; Adjusted for the baseline stratification factors: black versus non black, and cirrhosis versus no cirrhosis; Percent difference in SVR rates = 15.6, 95% CI 2-sided [6.5 to 24.8]

4. Secondary Outcome: Number of Participants Negative for HCV-RNA at FW 12
Description: Participants who had undetectable plasma HCV-RNA at FW 12. Also reported are participants for whom the HCV-RNA values were missing. 36 participant who switched over to Arm 8 from Arm 1, are included in the missing values for Arm 1.
  HCV-RNA in plasma samples was detected with an RT-PCR assay. The LLD for the assay was 29 IU/mL.
Time Frame: At FW 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm 1. PEG +RBV for 48 Wks (Part I) | Arm 2. PEG + RBV + BOC for 28 Wks (Part I) | Arm 3. PEG + RBV + BOC (From Wk 4) for 24 Wks (Part I) | Arm 4. PEG +RBV + BOC for 48 Wks (Part I) | Arm 5. PEG + RBV+ BOC (From Wk 4) for 44 Wks (Part I) | Arm 6. PEG + RBV + BOC for 48 Wks (Part II) | Arm 7. PEG +Low-dose RBV + BOC for 48 Wks (Part II)
Number analyzed (Participants) | 104 | 107 | 103 | 103 | 103 | 16 | 59
Participants
  HCV-RNA negative | 39 | 60 | 59 | 69 | 76 | 8 | 21
  Missing HCV-RNA at FW 12 | 42 | 13 | 11 | 12 | 14 | 2 | 17

5. Secondary Outcome: Number of Participants Negative for HCV-RNA at 72 Weeks Post Randomization
Description: Participants who had undetectable HCV-RNA at 72 weeks post randomization are reported. Participants with missing HCV-RNA values at 72 weeks post randomization are also reported.
  HCV-RNA in plasma samples was detected with an RT-PCR assay. The LLD for the assay was 29 IU/mL.
Time Frame: 72 weeks post randomization
Measure: Number; unit: Participants
Arm/Group | Arm 1. PEG +RBV for 48 Wks (Part I) | Arm 2. PEG + RBV + BOC for 28 Wks (Part I) | Arm 3. PEG + RBV + BOC (From Wk 4) for 24 Wks (Part I) | Arm 4. PEG +RBV + BOC for 48 Wks (Part I) | Arm 5. PEG + RBV+ BOC (From Wk 4) for 44 Wks (Part I) | Arm 6. PEG + RBV + BOC for 48 Wks (Part II) | Arm 7. PEG +Low-dose RBV + BOC for 48 Wks (Part II)
Number analyzed (Participants) | 104 | 107 | 103 | 103 | 103 | 16 | 59
Participants
  HCV-RNA negative | 38 | 53 | 56 | 67 | 76 | 8 | 20
  Missing HCV-RNA at 72 weeks post randomization | 45 | 25 | 18 | 17 | 20 | 6 | 22

6. Secondary Outcome: Number of Participants With an Early Virologic Response (EVR) That Achieved SVR
Description: Participants with undetectable HCV-RNA at TW 12 have EVR, and with undetectable HCV-RNA at FW 24 (up to EOF) achieved SVR.
  Participants missing data at FW 24 were considered to achieve SVR if
  1. he/she had undetectable HCV-RNA at FW 12 or later
  2. if he/she returned later to the study center and had undetectable HCV-RNA.
  HCV-RNA in plasma samples was detected with an RT-PCR assay. The LLD for the assay was 29 IU/mL.
Time Frame: At TW 12, and at FW 24 up to EOF
Population: Participants with an early virologic response (EVR).
Measure: Number; unit: Participants
Arm/Group | Arm 1. PEG +RBV for 48 Wks (Part I) | Arm 2. PEG + RBV + BOC for 28 Wks (Part I) | Arm 3. PEG + RBV + BOC (From Wk 4) for 24 Wks (Part I) | Arm 4. PEG +RBV + BOC for 48 Wks (Part I) | Arm 5. PEG + RBV+ BOC (From Wk 4) for 44 Wks (Part I) | Arm 6. PEG + RBV + BOC for 48 Wks (Part II) | Arm 7. PEG +Low-dose RBV + BOC for 48 Wks (Part II)
Number analyzed (Participants) | 37 | 85 | 85 | 81 | 85 | 11 | 35
Participants | 32 | 58 | 58 | 68 | 77 | 8 | 21

7. Secondary Outcome: Number of Participants With a Virologic Response at Follow-up Week 12 That Achieved SVR
Description: Treatment-naïve adults with CHC genotype 1 were assigned study medication. Participants with undetectable HCV-RNA at FW 12 that achieved SVR (have undetectable HCV-RNA at FW 24 (up to EOF) are reported.
  Participants missing data at FW 24 were considered to achieve SVR if
  1. he/she had undetectable HCV-RNA at FW 12 or later
  2. if he/she returned later to the study center and had undetectable HCV-RNA.
  HCV-RNA in plasma samples was detected with an RT-PCR assay. The LLD for the assay was 29 IU/mL.
Time Frame: At FW 12 and FW 24 up to EOF
Population: Participants with undetectable HCV-RNA at FW 12.
Measure: Number; unit: Participants
Arm/Group | Arm 1. PEG +RBV for 48 Wks (Part I) | Arm 2. PEG + RBV + BOC for 28 Wks (Part I) | Arm 3. PEG + RBV + BOC (From Wk 4) for 24 Wks (Part I) | Arm 4. PEG +RBV + BOC for 48 Wks (Part I) | Arm 5. PEG + RBV+ BOC (From Wk 4) for 44 Wks (Part I) | Arm 6. PEG + RBV + BOC for 48 Wks (Part II) | Arm 7. PEG +Low-dose RBV + BOC for 48 Wks (Part II)
Number analyzed (Participants) | 39 | 60 | 59 | 69 | 76 | 8 | 21
Participants
  HCV-RNA negative at EOF | 39 | 58 | 58 | 69 | 76 | 8 | 20
  HCV-RNA positive at EOF | 0 | 2 | 1 | 0 | 0 | 0 | 1
  Missing HCV-RNA at EOF | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With a Virologic Response at 72 Weeks Post Randomization That Achieved SVR
Description: Participants with undetectable HCV-RNA at 72 weeks post randomization that achieved SVR (have undetectable HCV-RNA at FW 24 up to EOF) are reported.
  Participants missing data at FW 24 were considered to achieve SVR if
  1. he/she had undetectable HCV-RNA at FW 12 or later
  2. if he/she returned later to the study center and had undetectable HCV-RNA.
  HCV-RNA in plasma samples was detected an the RT-PCR assay. The lower limit of detection (LLD) was 29 IU/mL.
Time Frame: At FW 24 up to EOF and at 72 weeks post randomization
Population: Participants who achieved SVR.
Measure: Number; unit: Participants
Arm/Group | Arm 1. PEG +RBV for 48 Wks (Part I) | Arm 2. PEG + RBV + BOC for 28 Wks (Part I) | Arm 3. PEG + RBV + BOC (From Wk 4) for 24 Wks (Part I) | Arm 4. PEG +RBV + BOC for 48 Wks (Part I) | Arm 5. PEG + RBV+ BOC (From Wk 4) for 44 Wks (Part I) | Arm 6. PEG + RBV + BOC for 48 Wks (Part II) | Arm 7. PEG +Low-dose RBV + BOC for 48 Wks (Part II)
Number analyzed (Participants) | 39 | 58 | 58 | 69 | 77 | 8 | 21
Participants
  HCV-RNA negative at 72 weeks post randomization | 38 | 53 | 56 | 67 | 76 | 8 | 20
  HCV-RNA positive at FW 24 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing HCV-RNA at 72 weeks post randomization | 1 | 5 | 2 | 2 | 1 | 0 | 1

ADVERSE EVENTS:
Groups:
- PEG +RBV for 48 Wks (Part I): Arm 1. PegIntron (1.5 μg/kg, once weekly [QW]) plus ribavirin (800 to 1400 mg/day) for 48 weeks.
  • Participants with detectable HCV-RNA levels after 24 weeks of treatment had the option of crossing over to receive 24 weeks of PegIntron, ribavirin, and boceprevir (800 mg, thrice a day [TID]) for 24 additional weeks. Total treatment duration was up to 54 weeks.
  Adverse events for 36 participants after they crossed over to Arm 8 are not included.
- PEG + RBV + BOC for 28 Wks (Part I): Arm 2. Boceprevir (800 mg TID) plus PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for up to 28 weeks.
- PEG + RBV + BOC (From Wk 4) for 24 Wks (Part I): Arm 3. PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for 4 weeks lead-in followed by boceprevir (800 mg TID) plus PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for up to 24 weeks.
- PEG +RBV + BOC for 48 Wks (Part I): Arm 4. Boceprevir (800 mg TID) plus PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for up to 48 weeks.
- PEG + RBV + BOC (From Wk 4) for 44 Wks (Part I): Arm 5. PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for 4 weeks lead-in followed by boceprevir (800 mg TID) plus PegIntron (1.5 μg/kg QW) and ribavirin (800 to 1400 mg/day) for up to 44 weeks.
- PEG + RBV + BOC for 48 Wks (Part II): Arm 6. PegIntron (1.5 μg/kg QW), ribavirin (800 to 1400 mg/day) and boceprevir (800 mg TID) for up to 48 weeks.
- PEG +Low-dose RBV + BOC for 48 Wks (Part II): Arm 7. PegIntron (1.5 μg/kg QW), ribavirin (400 to 1000 mg/day) and boceprevir (800 mg TID) for up to 48 weeks.
- PEG + RBV + BOC (From Wk 24) for 48 Wks (Part I): Arm 8. Participants that started in Arm 1 and had detectable HCV-RNA levels after 24 weeks of treatment had the option of receiving boceprevir (800 mg TID) with PegIntron (1.5 μg/kg QW), ribavirin (800 to 1400 mg/day). Participants that took the option of crossing over to receive 24 weeks of PegIntron, ribavirin, and boceprevir (800 mg TID) for 24 additional weeks constitute Arm 8. The total treatment duration was up to 54 weeks.
Arm/Group | PEG +RBV for 48 Wks (Part I) | PEG + RBV + BOC for 28 Wks (Part I) | PEG + RBV + BOC (From Wk 4) for 24 Wks (Part I) | PEG +RBV + BOC for 48 Wks (Part I) | PEG + RBV + BOC (From Wk 4) for 44 Wks (Part I) | PEG + RBV + BOC for 48 Wks (Part II) | PEG +Low-dose RBV + BOC for 48 Wks (Part II) | PEG + RBV + BOC (From Wk 24) for 48 Wks (Part I)
Serious Adverse Events (participants affected / at risk) | 8/104 | 10/107 | 8/103 | 10/103 | 6/103 | 1/16 | 3/59 | 2/36
Other Adverse Events (participants affected / at risk) | 102/104 | 106/107 | 102/103 | 103/103 | 102/103 | 16/16 | 59/59 | 29/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG +RBV for 48 Wks (Part I) (N=104) | PEG + RBV + BOC for 28 Wks (Part I) (N=107) | PEG + RBV + BOC (From Wk 4) for 24 Wks (Part I) (N=103) | PEG +RBV + BOC for 48 Wks (Part I) (N=103) | PEG + RBV + BOC (From Wk 4) for 44 Wks (Part I) (N=103) | PEG + RBV + BOC for 48 Wks (Part II) (N=16) | PEG +Low-dose RBV + BOC for 48 Wks (Part II) (N=59) | PEG + RBV + BOC (From Wk 24) for 48 Wks (Part I) (N=36)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERICARDITIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEAFNESS UNILATERAL (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIPLOPIA (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RETINAL ISCHAEMIA (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RETINOPATHY (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SCOTOMA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 0 (0) | 0 (0)
PERIODONTAL DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOCAL SWELLING (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MULTI-ORGAN FAILURE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CORNEAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERYSIPELAS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOBAR PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VULVAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANIMAL BITE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRUG TOXICITY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD AMYLASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LIPASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CERVICAL CORD COMPRESSION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IIIRD NERVE PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AGGRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALCOHOLISM (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEPENDENCE (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HOMICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANIC ATTACK (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PARANOIA (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UMBILICAL HERNIA REPAIR (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG +RBV for 48 Wks (Part I) (N=104) | PEG + RBV + BOC for 28 Wks (Part I) (N=107) | PEG + RBV + BOC (From Wk 4) for 24 Wks (Part I) (N=103) | PEG +RBV + BOC for 48 Wks (Part I) (N=103) | PEG + RBV + BOC (From Wk 4) for 44 Wks (Part I) (N=103) | PEG + RBV + BOC for 48 Wks (Part II) (N=16) | PEG +Low-dose RBV + BOC for 48 Wks (Part II) (N=59) | PEG + RBV + BOC (From Wk 24) for 48 Wks (Part I) (N=36)
ANAEMIA (Blood and lymphatic system disorders) | 35 (55) | 59 (96) | 55 (80) | 54 (79) | 58 (88) | 10 (22) | 14 (39) | 13 (13)
LEUKOPENIA (Blood and lymphatic system disorders) | 6 (15) | 7 (37) | 5 (12) | 5 (9) | 8 (12) | 1 (7) | 9 (58) | 1 (2)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 12 (32) | 23 (82) | 16 (30) | 26 (50) | 31 (71) | 2 (11) | 19 (88) | 8 (9)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 5 (7) | 1 (1) | 1 (1) | 6 (9) | 1 (1) | 5 (26) | 3 (3)
PALPITATIONS (Cardiac disorders) | 2 (3) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
TINNITUS (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 3 (3) | 7 (7) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 6 (6) | 2 (2) | 3 (3) | 1 (1) | 5 (9) | 1 (1) | 0 (0) | 0 (0)
CONJUNCTIVAL DISCOLOURATION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
CONJUNCTIVITIS (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
DRY EYE (Eye disorders) | 4 (4) | 1 (1) | 3 (4) | 6 (6) | 4 (4) | 2 (2) | 5 (5) | 0 (0)
EYE IRRITATION (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
RETINAL HAEMORRHAGE (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RETINOPATHY (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 7 (7) | 6 (6) | 2 (2) | 8 (8) | 7 (7) | 2 (2) | 3 (3) | 0 (0)
VISUAL IMPAIRMENT (Eye disorders) | 2 (2) | 1 (1) | 5 (5) | 7 (7) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 9 (12) | 4 (4) | 6 (6) | 10 (10) | 6 (7) | 1 (1) | 2 (3) | 2 (2)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5 (5) | 7 (8) | 5 (7) | 9 (9) | 12 (15) | 2 (2) | 5 (6) | 1 (1)
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 2 (2) | 2 (3) | 3 (4) | 4 (4) | 4 (4) | 2 (2) | 3 (3) | 0 (0)
CHEILITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 2 (2) | 1 (2) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 11 (13) | 5 (5) | 14 (17) | 9 (10) | 9 (10) | 1 (1) | 3 (3) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 23 (31) | 28 (40) | 27 (29) | 25 (30) | 29 (36) | 5 (5) | 14 (18) | 2 (2)
DRY MOUTH (Gastrointestinal disorders) | 5 (5) | 14 (15) | 8 (8) | 12 (15) | 10 (10) | 2 (2) | 5 (7) | 2 (3)
DYSPEPSIA (Gastrointestinal disorders) | 8 (9) | 6 (8) | 8 (8) | 9 (10) | 8 (8) | 1 (1) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 5 (5) | 11 (12) | 3 (4) | 8 (9) | 10 (11) | 1 (2) | 2 (2) | 1 (1)
GINGIVAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 7 (7) | 5 (6) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 45 (52) | 41 (50) | 42 (53) | 55 (80) | 48 (87) | 10 (13) | 35 (40) | 4 (4)
ORAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
PROCTALGIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
SALIVARY HYPERSECRETION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
STOMACH DISCOMFORT (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 2 (2) | 7 (8) | 5 (5) | 5 (7) | 4 (5) | 0 (0) | 0 (0) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 5 (7) | 24 (27) | 15 (21) | 25 (28) | 17 (23) | 7 (8) | 11 (14) | 2 (2)
ASTHENIA (General disorders) | 14 (18) | 9 (12) | 9 (18) | 20 (27) | 15 (26) | 1 (2) | 3 (3) | 3 (4)
CHEST DISCOMFORT (General disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
CHILLS (General disorders) | 35 (38) | 31 (39) | 31 (34) | 33 (37) | 35 (39) | 5 (6) | 26 (29) | 0 (0)
FATIGUE (General disorders) | 57 (62) | 65 (78) | 70 (80) | 51 (69) | 73 (95) | 11 (14) | 40 (55) | 5 (5)
IMPAIRED HEALING (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 25 (37) | 24 (26) | 21 (22) | 19 (20) | 15 (27) | 6 (6) | 11 (11) | 0 (0)
INJECTION SITE ERYTHEMA (General disorders) | 13 (13) | 9 (9) | 14 (14) | 7 (7) | 13 (13) | 1 (1) | 4 (4) | 1 (1)
INJECTION SITE RASH (General disorders) | 6 (6) | 3 (3) | 0 (0) | 3 (3) | 6 (6) | 1 (1) | 1 (1) | 0 (0)
INJECTION SITE REACTION (General disorders) | 10 (12) | 9 (9) | 5 (5) | 9 (9) | 11 (11) | 4 (4) | 21 (21) | 1 (1)
IRRITABILITY (General disorders) | 23 (23) | 25 (26) | 24 (27) | 15 (21) | 27 (32) | 3 (3) | 9 (11) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
PAIN (General disorders) | 8 (8) | 11 (11) | 9 (10) | 11 (12) | 5 (5) | 1 (1) | 11 (12) | 0 (0)
PYREXIA (General disorders) | 35 (55) | 27 (35) | 27 (34) | 40 (51) | 35 (53) | 7 (10) | 26 (31) | 0 (0)
TEMPERATURE INTOLERANCE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 3 (3) | 4 (6) | 1 (1) | 2 (2) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
EAR INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
EYE INFECTION (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 1 (1) | 3 (4) | 0 (0) | 3 (4) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
LARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (5) | 0 (0)
PHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (3) | 1 (1) | 1 (1) | 1 (1)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
RECTAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 3 (3) | 3 (4) | 3 (3) | 5 (7) | 5 (5) | 2 (3) | 1 (1) | 2 (2)
TINEA VERSICOLOUR (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 7 (7) | 1 (1) | 4 (4) | 7 (8) | 1 (1) | 6 (7) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 3 (4) | 3 (3) | 3 (3) | 2 (2) | 1 (2) | 1 (1) | 2 (2) | 0 (0)
BLOOD URIC ACID INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
HEART RATE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 9 (9) | 6 (6) | 8 (8) | 6 (8) | 9 (10) | 2 (2) | 8 (8) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 10 (11) | 10 (10) | 8 (8) | 13 (18) | 11 (15) | 2 (2) | 4 (5) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 12 (13) | 7 (7) | 14 (15) | 16 (18) | 12 (12) | 6 (6) | 16 (17) | 1 (1)
HYPERAMYLASAEMIA (Metabolism and nutrition disorders) | 1 (2) | 3 (4) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 3 (3) | 0 (0)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 21 (24) | 14 (20) | 22 (26) | 21 (25) | 19 (21) | 5 (7) | 11 (13) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5) | 7 (7) | 10 (13) | 9 (11) | 3 (3) | 5 (5) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 5 (7) | 4 (4) | 4 (4) | 6 (6) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 17 (17) | 31 (34) | 20 (20) | 21 (30) | 27 (33) | 4 (5) | 12 (15) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (4) | 0 (0) | 6 (7) | 4 (5) | 0 (0) | 2 (2) | 0 (0)
AMNESIA (Nervous system disorders) | 1 (1) | 1 (1) | 2 (3) | 5 (6) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 4 (5) | 7 (7) | 9 (9) | 7 (8) | 10 (11) | 0 (0) | 3 (4) | 0 (0)
DIZZINESS (Nervous system disorders) | 16 (18) | 19 (23) | 16 (18) | 21 (21) | 14 (18) | 7 (8) | 11 (16) | 2 (2)
DYSGEUSIA (Nervous system disorders) | 9 (10) | 23 (25) | 27 (28) | 33 (38) | 28 (31) | 7 (9) | 18 (20) | 7 (7)
HEADACHE (Nervous system disorders) | 45 (60) | 51 (66) | 41 (46) | 44 (52) | 54 (67) | 13 (13) | 29 (35) | 2 (2)
MEMORY IMPAIRMENT (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 5 (5) | 1 (1)
MIGRAINE (Nervous system disorders) | 2 (3) | 1 (1) | 2 (2) | 5 (5) | 3 (3) | 4 (6) | 1 (1) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 3 (4) | 5 (6) | 4 (4) | 6 (6) | 2 (2) | 1 (2) | 3 (3) | 0 (0)
SCIATICA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 3 (3) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 2 (3) | 4 (4) | 0 (0)
TRIGEMINAL NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 18 (21) | 16 (19) | 9 (10) | 15 (17) | 17 (20) | 1 (1) | 8 (11) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 22 (25) | 22 (29) | 20 (23) | 29 (34) | 20 (26) | 1 (1) | 14 (17) | 4 (5)
INSOMNIA (Psychiatric disorders) | 40 (50) | 36 (40) | 29 (37) | 40 (46) | 41 (48) | 7 (7) | 23 (27) | 7 (7)
MOOD SWINGS (Psychiatric disorders) | 2 (3) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
CHROMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
NOCTURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 1 (1) | 4 (4) | 6 (6) | 3 (3) | 6 (6) | 2 (2) | 5 (5) | 0 (0)
URETHRAL OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 5 (5) | 0 (0)
VULVOVAGINAL PRURITUS (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 20 (26) | 18 (27) | 22 (25) | 17 (21) | 19 (25) | 2 (2) | 8 (9) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 15 (20) | 18 (23) | 12 (12) | 16 (21) | 20 (25) | 4 (4) | 10 (14) | 2 (2)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6) | 2 (2) | 5 (6) | 11 (14) | 1 (1) | 4 (4) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4) | 2 (2) | 6 (7) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
INCREASED UPPER AIRWAY SECRETION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 11 (12) | 9 (10) | 5 (5) | 2 (2) | 2 (2) | 1 (1)
PARANASAL SINUS HYPERSECRETION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 0 (0) | 2 (2) | 4 (5) | 0 (0) | 3 (5) | 0 (0)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 3 (3) | 3 (3) | 4 (4) | 1 (1) | 2 (2) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 27 (28) | 36 (41) | 30 (34) | 30 (31) | 35 (38) | 5 (5) | 19 (19) | 2 (2)
DERMATITIS (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 1 (1) | 4 (5) | 1 (1) | 2 (4) | 2 (2) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 17 (17) | 12 (14) | 9 (10) | 22 (24) | 17 (18) | 3 (3) | 9 (13) | 4 (4)
ECZEMA (Skin and subcutaneous tissue disorders) | 4 (7) | 2 (2) | 7 (8) | 3 (4) | 4 (4) | 2 (2) | 2 (2) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 6 (6) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
INCREASED TENDENCY TO BRUISE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 16 (20) | 19 (23) | 19 (28) | 23 (35) | 19 (24) | 1 (1) | 11 (17) | 3 (3)
RASH (Skin and subcutaneous tissue disorders) | 6 (7) | 3 (5) | 6 (6) | 9 (12) | 9 (9) | 1 (1) | 1 (1) | 2 (2)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 2 (3) | 7 (9) | 5 (6) | 4 (9) | 3 (3) | 0 (0) | 2 (3) | 0 (0)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 6 (9) | 6 (7) | 0 (0) | 2 (3) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 5 (7) | 6 (7) | 1 (1) | 5 (5) | 4 (5) | 1 (1) | 8 (9) | 0 (0)
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 8 (10) | 9 (9) | 8 (9) | 17 (23) | 14 (17) | 1 (1) | 4 (6) | 0 (0)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 4 (4) | 1 (1) | 5 (6) | 1 (1) | 5 (7) | 1 (1)
SKIN LESION (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 2 (2)
URTICARIA (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 6 (6) | 2 (2) | 4 (4) | 1 (1) | 5 (5) | 0 (0) | 3 (4) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator agrees to provide to the sponsor thirty (30) days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication (including slides and texts of oral or other public presentations and texts of any transmission through any electronic media) that report any results of the study.